CLINICAL TRIAL: NCT04288076
Title: The Effect of Positive End Expiratory Pressure on Intracranial Pressure: The Brain and Lung Interaction (BALI) Study
Brief Title: The Brain and Lung Interaction (BALI) Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low eligibility rate
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Shahzad Shaefi, Assistant Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P000830
Record Dates: First submitted 2020-02-26; First posted 2020-02-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Intracranial Pressure; Mechanical Ventilation; Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEP Titration Arm (Experimental)
  Interventions: Other: PEEP Titrated Mechanical Ventilation

INTERVENTIONS:
Other: PEEP Titrated Mechanical Ventilation — Subjects will receive a sequential, step-wise increase in positive end-expired pressure from 5 cmH2O to 15 cmH2O and back down to 5 cmH20. Pleural pressure and intracranial pressure will be measured at each increment. PEEP will be increased by increments of 5 cmH2O. The physiologic measurements will be obtained at regular intervals (within 5 minutes at each PEEP level) throughout the PEEP titration period. The mode of mechanical ventilation (pressure or volume control), inspiratory time and fraction of inspired oxygen (FIO2) will be determined by the critical care team caring for the patient. In the event that PEEP is set > 5 cmH2O, measurements will be obtained from that starting point and increased to a maximum of 15 cmH2O. At the completion of the study patients will be returned to the PEEP level they were on prior to titration of the ventilator.

SUMMARY:
The purpose of this study is to understand the relationship between intracranial pressure and airway pressures during mechanical ventilation. This study is a single-center, prospective cohort study to be conducted at Beth Israel Deaconess Medical Center. The investigators will recruit patients with severe brain injury (GCS 8 or less) who receive intracranial pressure monitoring and mechanical ventilation as part of their routine medical care. The primary endpoint is the change in intracranial pressure as a function of positive end-expiratory pressure. There is only one study encounter with safety monitoring for up to 24 hours after. No additional follow up is required.

ELIGIBILITY:
Inclusion Criteria:

- Patients with severe brain injury (GCS 8 or less) who receive both mechanical ventilation and intracranial pressure monitoring as part of their standard medical care will be considered eligible.

Exclusion Criteria:

* Patients with esophageal varices
* Patients with esophageal trauma
* Patients with recent esophageal surgery
* Patients with coagulopathy (Platelets < 80k or INR> 2 )
* Other contraindication for esophageal manometry
* Patients who are receiving PEEP greater than 15 cmH2O within 24 hours prior to enrollment
* Intracranial hypertension (defined as ICP greater than 20 mmHg) within 48 hours prior to enrollment
* Decompressive hemi-craniectomy

Cessation Criteria: Study related ventilator adjustments and measurements will be stopped at any point during the intervention and ventilator settings will be returned to the pre-intervention settings under the following conditions:

* If ICP increases above 20mmHg, regardless of the duration of the event.
* If systolic blood pressure decreases below 90mmHg, regardless of the duration of the event.
* If systolic blood pressure increases above 180mmHg, regardless of the duration of the event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Change in intracranial pressure | Change from baseline to 20 minutes
  The primary endpoint is the change in intracranial pressure as a function of positive end-expiratory pressure.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rincon F, Ghosh S, Dey S, Maltenfort M, Vibbert M, Urtecho J, McBride W, Moussouttas M, Bell R, Ratliff JK, Jallo J. Impact of acute lung injury and acute respiratory distress syndrome after traumatic brain injury in the United States. Neurosurgery. 2012 Oct;71(4):795-803. doi: 10.1227/NEU.0b013e3182672ae5. PMID 22855028
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Malhotra A. Low-tidal-volume ventilation in the acute respiratory distress syndrome. N Engl J Med. 2007 Sep 13;357(11):1113-20. doi: 10.1056/NEJMct074213. PMID 17855672
- [Background] Quilez ME, Fuster G, Villar J, Flores C, Marti-Sistac O, Blanch L, Lopez-Aguilar J. Erratum to: Injurious mechanical ventilation affects neuronal activation in ventilated rats. Crit Care. 2015 Oct 27;19:379. doi: 10.1186/s13054-015-1076-5. No abstract available. PMID 26506991
- [Background] Pelosi P, Rocco PR. The lung and the brain: a dangerous cross-talk. Crit Care. 2011;15(3):168. doi: 10.1186/cc10259. Epub 2011 Jun 30. PMID 21722336
- [Background] Pelosi P, Ferguson ND, Frutos-Vivar F, Anzueto A, Putensen C, Raymondos K, Apezteguia C, Desmery P, Hurtado J, Abroug F, Elizalde J, Tomicic V, Cakar N, Gonzalez M, Arabi Y, Moreno R, Esteban A; Ventila Study Group. Management and outcome of mechanically ventilated neurologic patients. Crit Care Med. 2011 Jun;39(6):1482-92. doi: 10.1097/CCM.0b013e31821209a8. PMID 21378554
- [Background] Stevens RD, Lazaridis C, Chalela JA. The role of mechanical ventilation in acute brain injury. Neurol Clin. 2008 May;26(2):543-63, x. doi: 10.1016/j.ncl.2008.03.014. PMID 18514826
- [Background] Caricato A, Conti G, Della Corte F, Mancino A, Santilli F, Sandroni C, Proietti R, Antonelli M. Effects of PEEP on the intracranial system of patients with head injury and subarachnoid hemorrhage: the role of respiratory system compliance. J Trauma. 2005 Mar;58(3):571-6. doi: 10.1097/01.ta.0000152806.19198.db. PMID 15761353
- [Background] Huynh T, Messer M, Sing RF, Miles W, Jacobs DG, Thomason MH. Positive end-expiratory pressure alters intracranial and cerebral perfusion pressure in severe traumatic brain injury. J Trauma. 2002 Sep;53(3):488-92; discussion 492-3. doi: 10.1097/00005373-200209000-00016. PMID 12352486
- [Background] Mascia L, Grasso S, Fiore T, Bruno F, Berardino M, Ducati A. Cerebro-pulmonary interactions during the application of low levels of positive end-expiratory pressure. Intensive Care Med. 2005 Mar;31(3):373-9. doi: 10.1007/s00134-004-2491-2. Epub 2005 Jan 25. PMID 15668765